CLINICAL TRIAL: NCT05587556
Title: Analysis of Clinical Outcomes and Complications in Patients Received Liver Transplantation: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Long-Bin Jeng, Professor, China Medical University Hospital
Other Study IDs: CMUH110-REC1-235
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-01

CONDITIONS: Liver Transplant, Liver Cancer, Immunosuppressant
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplantation is the last-line method for liver failure. Thomas Starzl completed the first liver transplant in 1967, liver transplantation is developing rapidly. In Taiwan, the first liver transplantation was started in 1984, and the living donor liver transplantation was started in 1994. According to statistics from the Taiwan Organ Transplant Registration Center, from 2005 to 2018, a total of 6,211 liver transplants were completed in Taiwan, and the three-year survival rate was 78.9%.

The success rate of liver transplantation is closely related to the operation method, complications, the patient's conditions, and postoperative care. Besides, Liver cancer is the sixth most common cancer in the whole world and also the fourth leading cause of cancer-related death. Approximately 90% of patients are diagnosed with liver cirrhosis at the same time when they are diagnosed with liver cancer. Once the late stages of liver cirrhosis happen, the effect of treatment will be reduced. Therefore, liver transplantation is the only treatment option that can solve the simultaneous occurrence of liver cirrhosis and liver cancer. Since 1996, liver transplantation has been used to treat liver cancer, the organ source is always the Achilles tendon of organ transplantation. Therefore, Milan criteria was designed to achieve the justice of organ share. However, living donor liver transplant is more popular in Eastern countries because of religious factors and ethical issues and many famous medical centers are trying to expand the original Milan or UCSF criteria, such as Kyoto criteria and Up-to-7 criteria, hoping to save more patients. However, with the expansion of conditions, the chance of recurrence or metastasis after transplantation is bound to increase. According to reports from different famous medical centers, the recurrence rate of liver cancer after liver transplantation is about 10-20%.

Therefore, we assume that patients with liver replacement caused by different diseases may have other postoperative conditions and complications. This study will review the preoperative diagnosis, surgical status, postoperative status, medication status, complications and recurrence of liver transplant patients in our hospital for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1400 patients who received liver transplantation or patients who were followed up after liver transplantation

Exclusion Criteria:

* Patients who do not meet the inclusion and exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preoperative diagnosis, surgical status, postoperative status, presence or absence of complications, postoperative medication status, medication complications and post-recurrence treatment for patients who received liver transplantation or who were followed up after liver transplantation difference analysis
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The survial rate of the patients | Jan. 2002 to Dec. 2021
  To investigate whether preoperative diagnosis, surgical status, postoperative status, medication status, complications and recurrence have significant differences in the survival rate of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Long-Bin Jeng, Principal Investigator — Organ Transplantation Center, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan